CLINICAL TRIAL: NCT05517161
Title: Roll for Intervention - a Critical Look at the Practicability of Table-top Roll Playing Games as Communication Intervention for Traumatic Brain Injury
Brief Title: Roll for Intervention - TBI Group Treatment
Status: Completed | Type: Observational
Sponsor: Moravian University (Other)
Responsible Party: Principal Investigator, Louise Keegan, Associate Professor & Program Director of Speech-Language Pathology, Moravian University
Other Study IDs: 22-015
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Communication Disorder, Social
MeSH Terms: conditions — Social Communication Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with TBI
  Interventions: Behavioral: INSIGHT

INTERVENTIONS:
Behavioral: INSIGHT — See Keegan et al., 2020

SUMMARY:
Communication group intervention for individuals with Traumatic Brain Injury based on INSIGHT protocol (Keegan et al, 2020) with roll playing game focus

DETAILED DESCRIPTION:
Individuals with TBI recruited to participate in a study about applying INSIGHT protocol to a virtual roll playing game environment. The game 'monsters of the week' will be used to administer the cognitive-communication ingredients outlined by INSIGHT (Keegan et al 2020) and progress towards social communication goals will be documented throughout the course of participating in the roll playing campaign (7-8 weeks - meeting 2 hours each week). The individuals without neurological disorders will follow the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe TBI more than 1 year ago

Exclusion Criteria:

* other neurological diagnoses prior to TBI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: individuals who have received a brain injury at least 1 year prior to enrollment.
  Group 2: age, education and gender matched individuals who have no history of neurological difficulties
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Goal Attainament Scaling - change over time | Week 2, 3,4,5,6,7, 8 and 9 of the 10week study protocol
  Assessing change over time on five point scaled goals - goal rated each week for 8 weeks.

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status Update | During week 1 and week 10 of the 10 week protocol
  Randolf (2012) standardized norm referenced assessment measure of cognitive skills (memory and attention etc.)
Functional Assessment of Verbal Reasoning and Executive Strategies | During week 1 and week 10 of the 10 week protocol
  MacDonald (2005) standardized norm referenced assessment measure of problem solving and reasoning
Sydney psychosocial reintegration scale version 2 (SPRS-2) | During week 1 and week 10 of the 10 week protocol
  Tate (2012) standardized likert based questionnaire (12, 1-5 ratings, where higher scores = better performance)
Satisfaction with life scale (SWLS) | During week 1 and week 10 of the 10 week protocol
  Diener et al (1985), likert measurement scale questionnaire, 5 1-7 ratings, higher scores = better performance
Latrobe Communication Questionnaire (LCQ) | During week 1 and week 10 of the 10 week protocol
  Douglas et al (2000), likert measurement scale questionnaire, 30 1-4 ratings, higher scores = better performance

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Keegan, Principal Investigator — Moravian University
Locations (1):
- Moravian University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No